CLINICAL TRIAL: NCT04120961
Title: Safety and Efficacy of Prolonged Use of Bivalirudin 4 Hours After Elective PCI in Patients With CHD (COBER Study)
Brief Title: Safety and Efficacy of Prolonged Use of Bivalirudin 4 Hours After ePCI (COBER Study)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: KY20190823-05
Record Dates: First submitted 2019-09-29; First posted 2019-10-09 (Actual); Last update posted 2022-08-09 (Actual); Status verified 2022-08

CONDITIONS: Coronary Heart Disease
Keywords: bivalirudin; prolonged use; peri-operative myocardial injury; percutaneous coronary intervention
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- prolonged continuous use of bivalirudine (Experimental): A total of 165 patients are assigned to group with prolonged continuous use of bivalirudin after randomization schedule.
  Interventions: Drug: prolonged continuous use of bivalirudin
- bivalirudin use during ePCI (Other): A total of 165 patients are assigned to group with bivalirudin use during ePCI after randomization schedule.
  Interventions: Drug: bivalirudin use during ePCI

INTERVENTIONS:
Drug: prolonged continuous use of bivalirudin — prolonged continuous use of bivalirudin 4 hours after elective PCI (dose: 0.75 mg/kg bolus plus 1.75 mg/kg per hour)
  Other Names: prolonged continuous use of bivalirudin 4 hours after elective PCI
  Arms: prolonged continuous use of bivalirudine
Drug: bivalirudin use during ePCI — bivalirudin use during ePCI (0.75 mg/kg bolus plus 1.75 mg/kg per hour)
  Other Names: bivalirudin use during ePCI period
  Arms: bivalirudin use during ePCI

SUMMARY:
Since the development of percutaneous coronary intervention (PCI) in patients with coronary heart disease (CHD), unfractionated heparin (UFH) and low molecular weight heparin (LWMH) have been the preferred anticoagulants in peri-operative period. However, UFH has some defects, such as incomplete and unstable inhibition of thrombin, large individual differences, multiple monitoring of activated coagulation time (ACT), ineffective thrombin binding to fibrin, non-specific protein binding and induced thrombocytopenia (HIT). Compared with UFH, LWMH has lower non-specific protein binding rate, but it is not superior to UFH in efficacy, hemorrhage and HIT.

Bivalirudin can bind specifically to thrombin catalytic site and anionic external binding site, directly inhibit thrombin activity, thereby inhibiting thrombin-catalyzed and induced reactions. At the same time, thrombin can also inactivate it by enzymatic hydrolysis of bivalirudin. Therefore, the inhibition of bivalirudin on thrombin is reversible and transient, and the risk of bleeding after drug withdrawal is relative small. It has been reported that bivalirudin can significantly reduce the risk of peri-operative bleeding during PCI period compared with UFH. Clopidogrel had not yet played a role in most patients after emergency PCI, and there was a "blank period" for 2-4 hours without effective antithrombotic concentration, which was also the peak period of acute stent thrombosis. Han and coworkers have shown that for acute myocardial infarction (AMI) patients undergoing emergency PCI, whether or not glycoprotein IIb/IIIa inhibitors were added, prolonged peri-operative use of bivalrudin was significantly better than UFH in terms of net clinical adverse event. However, for patients with elective PCI (ePCI), prolonged bivalirudin use was only used in some patients in REPLACE-2 and ISAR-REACT-3 studies, and the prolonged time of bivalrudin use after ePCI was not definite.

Therefore, in the current study we aim to explore the efficacy and safety of prolonged bivalirudin use 4 hours after elective PCI in patients with CHD.

DETAILED DESCRIPTION:
The current study is designed as a single-center, randomized and prospective study aiming to evaluate the safety and efficacy of prolonged continuous use of bivalirudin 4 hours after ePCI for the treatment of peri-operative myocardial injury (PMI) compared with the bivalirudin use during ePCI. Based on previous study reported and estimated 10% loss follow-up of these patients in each arm, a total of 330 patients with CHD were required in our study, and with 165 patients per group as a ratio of 1:1 randomization.

ELIGIBILITY:
Inclusion Criteria:

* De novo lesions
* elective PCI
* Only single coronary artery treated at this time

Exclusion Criteria:

* Those who meet the diagnostic criteria of acute myocardial infarction
* Patients with cardio-genic shock
* Patients with multiple organ failure
* Patients allergic to contrast
* Patients who can not tolerate dual antiplatelet therapy
* Patients who can't tolerate anticoagulation
* Recently infected patients
* Patients with hepatorenal dysfunction
* Thrombotic lesion of coronary artery
* Chronic total coronary occlusion lesion
* Patients with complex coronary bifurcation requiring two stent strategy
* Severe coronary calcified lesion
* Patients with percutaneous coronary angioplasty
* Patients with directional coronary atherectomy or rotational atherectomy
* Patients with drug coated balloon treatment
* Patients with bioabsorbable vascular scaffold implantation
* Previous percutaneous coronary intervention
* Previous coronary artery bypass graft
* Patients with active stage of autoimmune disease

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Actual)
Dates: Start 2019-09-20 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
The incidence rate of PMI in CHD patients 3 days after ePCI | Clinical follow up at 3 days after ePCI
  the incidence rate of PMI indicated by the changes of myocardial injury biomarkers (such as TNI and CK-MB) in CHD patients between prolonged use of bivalirudin and bivalirudin use during ePCI groups

SECONDARY OUTCOMES:
The incidence rate of MACEs and bleeding | Clinical follow up at 7 days after ePCI
  The incidence rate of major adverse cardiac events and bleeding between prolonged use of bivalirudin and bivalirudin use during ePCI groups

CONTACTS AND LOCATIONS:
Overall Officials: Zhiming Wu, MD, Principal Investigator — Nanjing First Hospital, Nanjing Medical University
Locations (1):
- Nanjing First Hospital, Nanjing Medical University, Nanjing, Jiangsu, China

REFERENCES:
- [Background] Han Y, Guo J, Zheng Y, Zang H, Su X, Wang Y, Chen S, Jiang T, Yang P, Chen J, Jiang D, Jing Q, Liang Z, Liu H, Zhao X, Li J, Li Y, Xu B, Stone GW; BRIGHT Investigators. Bivalirudin vs heparin with or without tirofiban during primary percutaneous coronary intervention in acute myocardial infarction: the BRIGHT randomized clinical trial. JAMA. 2015 Apr 7;313(13):1336-46. doi: 10.1001/jama.2015.2323. PMID 25775052
- [Background] Lincoff AM, Bittl JA, Harrington RA, Feit F, Kleiman NS, Jackman JD, Sarembock IJ, Cohen DJ, Spriggs D, Ebrahimi R, Keren G, Carr J, Cohen EA, Betriu A, Desmet W, Kereiakes DJ, Rutsch W, Wilcox RG, de Feyter PJ, Vahanian A, Topol EJ; REPLACE-2 Investigators. Bivalirudin and provisional glycoprotein IIb/IIIa blockade compared with heparin and planned glycoprotein IIb/IIIa blockade during percutaneous coronary intervention: REPLACE-2 randomized trial. JAMA. 2003 Feb 19;289(7):853-63. doi: 10.1001/jama.289.7.853. PMID 12588269
- [Background] Schulz S, Mehilli J, Ndrepepa G, Neumann FJ, Birkmeier KA, Kufner S, Richardt G, Berger PB, Schomig A, Kastrati A; Intracoronary Stenting and Antithrombotic Regimen: Rapid Early Action for Coronary Treatment (ISAR-REACT) 3 Trial Investigators. Bivalirudin vs. unfractionated heparin during percutaneous coronary interventions in patients with stable and unstable angina pectoris: 1-year results of the ISAR-REACT 3 trial. Eur Heart J. 2010 Mar;31(5):582-7. doi: 10.1093/eurheartj/ehq008. Epub 2010 Feb 11. PMID 20150324
- [Background] Devereaux PJ, Xavier D, Pogue J, Guyatt G, Sigamani A, Garutti I, Leslie K, Rao-Melacini P, Chrolavicius S, Yang H, Macdonald C, Avezum A, Lanthier L, Hu W, Yusuf S; POISE (PeriOperative ISchemic Evaluation) Investigators. Characteristics and short-term prognosis of perioperative myocardial infarction in patients undergoing noncardiac surgery: a cohort study. Ann Intern Med. 2011 Apr 19;154(8):523-8. doi: 10.7326/0003-4819-154-8-201104190-00003. PMID 21502650
- [Derived] Wu Z, Meng P, Guo Y, You W, Wu X, Ye F. Prolonged infusion of bivalirudin after elective percutaneous coronary intervention protects against procedural myocardial injury (a COBER study)-a randomized trial. Sci Rep. 2023 Apr 24;13(1):6667. doi: 10.1038/s41598-023-34008-y. PMID 37095298